CLINICAL TRIAL: NCT01773083
Title: Randomized Controlled Trial Investigating the Efficacy and Safety of Nebulized Heparin Versus Placebo in Burn Patients With Inhalation Trauma (Hepburn)
Brief Title: Trial of Nebulized Heparin Versus Placebo for Inhalation Trauma
Acronym: Hepburn
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment of patients and high costs associated with the purchase and blinding of study medication
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Burns Foundation (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof. Dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HepBurn; 2012-003289-42 (EudraCT Number)
Record Dates: First submitted 2013-01-16; First posted 2013-01-23 (Estimated); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Inhalation Injury; Burn Injury
Keywords: Inhalation trauma; pulmonary coagulopathy; heparin nebulization; mechanical ventilation
MeSH Terms: conditions — Burns | interventions — Heparin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- unfractionated heparin (Experimental): 25.000 IU/5 ml, will be nebulized 4 hourly (i.e. 6 times daily)
  Interventions: Drug: unfractionated heparin
- placebo (Placebo Comparator): Sterile sodium chloride (NaCl 0.9%, Pfizer), in 5 ml, will be nebulized every 4 hours (i.e. 6 times daily)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: unfractionated heparin — nebulized 6 times daily, daily dose 150.000 IU for the maximum duration of 14 days
  Other Names: unfractionated heparin sodium, EV Product Code: SUB02475MIG,; Marketing Authorisation number: RVG 01372; ATC codes: B01AB01
  Arms: unfractionated heparin
Drug: placebo — Placebo: Sterile saline nebulized 6 times daily for the maximum duration of 14 days
  Other Names: sterile sodium chloride (NaCl 0.9%)
  Arms: placebo

SUMMARY:
The purpose of this international multi-center double-blind randomized placebo-controlled trial is to determine the effect of nebulized heparin, compared to placebo, on the number of ventilator-free days at day 28, in burn patients with confirmed inhalation trauma requiring mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age > 18 years
* Need for invasive mechanical ventilation
* Confirmed inhalation trauma (bronchoscopically)

Exclusion Criteria:

* > 36 hours after trauma
* Receiving invasive ventilation > 24 hours
* Expected duration of mechanical ventilation < 24 hours
* Chronic obstructive pulmonary disease GOLD stage III and IV
* Any history of pulmonary hemorrhage in the past 3 months
* Any history of significant bleeding disorder
* Known allergy to heparin, including heparin-induced thrombocytopenia
* Pregnancy or breast feeding
* Unlikely to survive for > 72 hours
* Total body surface area (TBSA) > 60%
* Witnessed or proven aspiration (i.e., confirmed by bronchoscopy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Number of ventilator-free days at day 28 | at day 28
  The number of ventilator-free days is defined as the number of days a patient is breathing without assist of a ventilator during the first 28 days; thus, the patient must be free of mechanical ventilation for 24 hours to have one ventilator-free day; if after successful detubation the patient requires a reintubation due to a surgical procedure, this reintubation will not count as a ventilator day - however, the day(s) will be counted as ventilator day(s) if mechanical ventilation is prolonged after surgery due to respiratory insufficiency.

SECONDARY OUTCOMES:
Clinical outcome parameters | daily or at day 28 and day 90
  Clinical outcome parameters will include but not be restricted to: (a) length of stay (ICU and hospital); (b) mortality (28- and 90 days); (c) mortality (ICU and hospital); (d) daily Lung Injury Score (LIS); (e) daily Oxygenation Index (OI) ; (f) daily Sequential Organ Failure Assessment (SOFA)-scores ; (g) cumulative dosages of sedatives; (h) incidence of Ventilator-associated Pneumonia (VAP); (i) total number of bronchoscopy-guided cleaning of the larger airway
Laboratory outcome parameters | Blood and lavage samples: on admission day and every other day for a maximum period of 14 days
  Levels of markers of coagulation and fibrinolysis in blood and lung lavage fluid, Levels of markers of inflammation in blood and lung lavage fluid, Biomarkers of lung injury in blood and lung lavage fluid
Safety parameters | daily, for a maximum period of 28 days
  Safety parameters will include but not be restricted to: Occurrence of serious bleedings, any other transfusion of blood products - red cells and/or platelets and/or plasma, Confirmed Heparin induced thrombocytopenia, prolonged activated partial thromboplastin time (aPTT > 150 seconds)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus J Schultz, MD-PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (8):
- St Vincent's Hospital, Melbourne, Victoria, Australia
- Belgium (3):
  - University Hospital, Gent, Ghent, Oost-Vlaanderen
  - University Hospital Gasthuisberg - Leuven, Leuven, Vlaams-Brabant
  - Ziekenhuis Netwerk Antwerpen- Stuivenberg, Antwerp
- Netherlands (4):
  - Academic Medical Center, Amsterdam, North Holland
  - Red Cross Hospital, Beverwijk, the Netherlands, Beverwijk, North Holland
  - Maasstad Hospital, Rotterdam, South Holland
  - Martini Hospital, Groningen

REFERENCES:
- [Derived] Glas GJ, Muller J, Binnekade JM, Cleffken B, Colpaert K, Dixon B, Juffermans NP, Knape P, Levi MM, Loef BG, Mackie DP, Malbrain M, Schultz MJ, van der Sluijs KF. HEPBURN - investigating the efficacy and safety of nebulized heparin versus placebo in burn patients with inhalation trauma: study protocol for a multi-center randomized controlled trial. Trials. 2014 Mar 25;15:91. doi: 10.1186/1745-6215-15-91. PMID 24661817
- See also: HEPBURN website — https://sites.google.com/site/hepburnstudy/